CLINICAL TRIAL: NCT03890354
Title: Robot-Assisted or Laparoscopic Resection for Gastric Subepithelial Tumor With Hand-Sewn Repair, a Case Series
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/1006
Record Dates: First submitted 2019-03-24; First posted 2019-03-26 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Gastric Mass
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hand-Sewn Repair — gastotomy to identify and remove gastric subepithelium tumor and hand sawn repair

SUMMARY:
There are a lot of surgical techniques in minimally-invasive surgery to remove gastric subepithelium tumor. Surgical approach depend on location and size of tumor. Usefully used Endostapler to cut stomach include lesion. For tumors in difficult locations some surgeons prefer laparoscopic and endoscopic cooperation or use the intragastric port technique to identify and remove the mass. But in complex procedures, gastotomy and hand sawn to identify and remove gastric subepithelium tumor is a simple technique and easy to apply. This study demonstrates the safety and effectiveness of this technique.

DETAILED DESCRIPTION:
: A retrospective chart review was made of all patients who presented with gastric subepithelial tumor and underwent laparoscopic or robotic resection at Ramathibodi Hospital during 2012-2018. Surgical outcomes and complication of gastotomy and hand-sewn repair were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* all patients who presented with gastric subepithelial tumor and underwent laparoscopic or robotic resection at Ramathibodi Hospital during 2012-2018.

Exclusion Criteria:

* conversion to open surgery

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients who presented with gastric subepithelial tumor and underwent laparoscopic or robotic resection
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Post operative complication | 7 day
  anastomosis leak
Post operative compliction | 7 day
  wound infection

SECONDARY OUTCOMES:
Surgical outcome | 7 day
  Complete remove mass with out rupture

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi Hospital
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No